CLINICAL TRIAL: NCT06435923
Title: A Phase 1, Open-Label Trial to Assess the Absorption, Metabolism, Excretion, and Mass Balance of [14C]-Darigabat Following a Single Oral Dose in Healthy Adult Male Participants
Brief Title: A Trial to Assess the Absorption, Metabolism, Excretion, and Mass Balance of [14C]-Darigabat After a Single Oral Dose in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-865-HV-1004
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants
MeSH Terms: interventions — PF-06372865

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Darigabat (Experimental): Participants will receive a single oral dose of darigabat.
  Interventions: Drug: [14C]-darigabat

INTERVENTIONS:
Drug: [14C]-darigabat — Oral capsule
  Other Names: CVL-865; PF-06372865

SUMMARY:
The primary purpose of this trial is to determine the mass balance, routes, and rates of elimination of total radioactivity and characterize the pharmacokinetics (PK) of darigabat, and total radioactivity in plasma and whole blood following administration of a single oral dose of [14C]-darigabat in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index of 18.5 to 35.0 kilograms per square meters (kg/m^2), inclusive, and a total body weight ≥50 kg [110 Pounds (lbs)] at Screening.
2. A male participant who is sexually active with a pregnant or a nonpregnant partner of childbearing potential must agree to use a condom during the trial and for 93 days after the dose of investigational medicinal product (IMP). In addition, male participants should not donate sperm for a minimum of 93 days following the dose of IMP.
3. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus, thyroid disorders), malignancy, hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
2. "Yes" responses for any of the following items on the Columbia-Suicide Severity Rating Scale (C-SSRS) (within the individual's lifetime):

   * Suicidal Ideation Item 3 (Active Suicidal Ideation with Any Methods [Not Plan] without Intent to Act)
   * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan)
   * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent)
   * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior) "Yes" responses for any of the following items on the C-SSRS (within past 12 months):
   * Suicidal Ideation Item 1 (Wish to be Dead)
   * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts) Serious risk of suicide in the opinion of the investigator is also exclusionary.
3. Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, and cholecystectomy.
4. Positive result for human immunodeficiency viruses (HIV) antibody, hepatitis B surface antigen, hepatitis B total core antibody, or hepatitis C antibody with detectable viral Ribonucleic acid (RNA) levels at Screening. Note: Positive or indeterminate test result for hepatitis C antibody should follow with hepatitis C virus polymerase chain reaction (PCR) RNA test. If result is positive, the participant is excluded.
5. Positive drug screen [including cotinine and Tetrahydrocannabinol (THC)] or a positive test for alcohol.
6. Known allergy or hypersensitivity to the IMP, closely related compounds, or any of their specified ingredients.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — U.S. Food and Drug Administration (FDA) recommends that radiation exposure to participants should be kept as low as is reasonably achievable, and there is no available data to suggest metabolism of the darigabat is different in women versus men. Hence, female participants are excluded from this study.
Enrollment: 8 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Time Curve (AUC) from Time Zero to Infinity (AUCinf) of Darigabat | Pre-dose and at multiple time points post-dose up to Day 15
AUC from Time 0 to the Time of the Last Measured Concentration (AUClast) of Darigabat | Pre-dose and at multiple time points post-dose up to Day 15
Maximum Observed Plasma Concentration (Cmax) of Darigabat | Pre-dose and at multiple time points post-dose up to Day 15
Time to Last Quantifiable (Tlast) Concentration of Darigabat | Pre-dose and at multiple time points post-dose up to Day 15
Time to Maximum Observed Concentration (Tmax) of Darigabat | Pre-dose and at multiple time points post-dose up to Day 15
Terminal Phase Half-life (t½) of Darigabat | Pre-dose and at multiple time points post-dose up to Day 15
Apparent Total Clearance After Oral Administration (CL/F) of Darigabat | Pre-dose and at multiple time points post-dose up to Day 15
Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Darigabat | Pre-dose and at multiple time points post-dose up to Day 15
Ratio of Plasma AUCinf for Darigabat to Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Ratio of Whole Blood AUCinf for Total Radioactivity to Plasma Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
Amount Excreted in Urine (Aeu) of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
  Urine PK parameters will be assessed.
Amount Excreted in Feces (Aef) of Total Radioactivity | Pre-dose and at multiple time points post-dose up to Day 15
  Fecal PK parameters will be assessed.

SECONDARY OUTCOMES:
Metabolite Profile of [14C]-darigabat in Plasma, Urine and Feces | Pre-dose and at multiple time points post-dose up to Day 15
Identification of [14C]-darigabat Metabolites Found in Plasma, Urine and Feces | Pre-dose and at multiple time points post-dose up to Day 15
Structural Elucidation of [14C]-darigabat Metabolites ≥10% of the Total [14C]-darigabat Radioactivity Found in Plasma, Urine and Feces | Pre-dose and at multiple time points post-dose up to Day 15
Number of Participants with Adverse Events (AEs) | Up to Day 16
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to Day 15
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 15
Number of Participants with Clinically Significant Changes in Laboratory Assessments | Up to Day 15
Number of Participants with Clinically Significant Changes in Physical and Neurological Examination Results | Up to Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No